CLINICAL TRIAL: NCT01148888
Title: The Effect of Magnesium Sulfate on Motor and Somatosensory Evoked Potentials in Children Undergoing Scoliosis Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mark Crawford, Anesthesiologist-In-Chief, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000014574
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Scoliosis
Keywords: pediatrics; Anaesthesia; Scoliosis; Magnesium
MeSH Terms: conditions — Scoliosis | interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnesium Sulfate (Experimental): The study will be conducted in the 45 minute interval between the completion of spinal instrumentation and the completion of skin closure. Once the spinal instrumentation is complete and the integrity of the spinal cord pathways is confirmed using SEPs and MEPs, magnesium will be administered for the remainder of surgery.
  Interventions: Drug: Magnesium

INTERVENTIONS:
Drug: Magnesium — Magnesium will be administered intravenously at a dose of 50 mg/kg bolus followed by an infusion of 10 mg/kg/hr.

SUMMARY:
The primary objective of this study is to determine whether magnesium sulfate has a clinically important effect on the amplitude and latency of somatosensory and motor evoked potentials in patients undergoing surgical correction of idiopathic scoliosis.

DETAILED DESCRIPTION:
Motor and somatosensory evoked potentials are continuously monitored in the setting of scoliosis surgery to evaluate the integrity of spinal cord pathways. Detection of neural irritation or injury using motor or somatosensory evoked potentials allows the surgeon to modify technique to reverse the insult and proceed without spinal cord compromise. To facilitate evoked potential monitoring, anesthetic agents that attenuate the evoked responses must be avoided.Several different agents have been studied to try to diminish the acute opioid tolerance and/or hyperalgesia seen with remifentanil.

Two studies investigated the effect of magnesium sulfate on intraoperative remifentanil-induced hyperalgesia. In both studies, post-operative pain scores and opioid consumption were decreased in those patients who received magnesium.

Our aim is to establish that magnesium sulfate does not adversely affect somatosensory evoked potentials (SEPs) and motor evoked potentials (MEPs) in patients undergoing correction of idiopathic scoliosis. Future clinical trials can then be performed investigating the effect of magnesium sulfate on remifentanil-induced hyperalgesia in the same population.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status I or II
* Adolescent children aged 12 to 18 years undergoing surgery for idiopathic scoliosis

Exclusion Criteria:

* Magnesium use within the last two weeks, either intravenous or oral supplements
* Patients with known electrolyte imbalances or conduction disorders. (Sodium <135 or >143 mmol/L OR Potassium < 3.7 or > 5.0 mmol/L if 12 to 15 yrs; Potassium <3.7 or >4.8 mmol/L if 16 to 18 yrs)
* Renal, cardiac or neuromuscular disorders.(Urea < 2.9 or > 7.1 mmol/L OR Creatinine >79 µmol/L if < 13 yrs; Creatinine > 98 µmol/L if >= 14 yrs)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Somatosensory and motor evoked potentials | Baseline
  Cortical SEPs will be measured from Cz-Fpz or Ci-Cc (10-20 system of head measurement) and the amplitudes will be taken from the first positive deflection to first negative deflection (P1-N1) after supramaximal stimulation of the posterior tibial nerves at the medial malleolus. The MEP peak-to-peak amplitudes will be measured from left and right tibialis anterior and abductor hallucis muscles. Stimulation parameters will be varied in order to achieve the maximum amplitude values. Evoked potentials will be measured before and at 10 and 30 minutes after the start of the magnesium infusion.
Somatosensory and motor evoked potentials | 10 and 30 minutes after the start of the magnesium infusion
  Cortical SEPs will be measured from Cz-Fpz or Ci-Cc (10-20 system of head measurement) and the amplitudes will be taken from the first positive deflection to first negative deflection (P1-N1) after supramaximal stimulation of the posterior tibial nerves at the medial malleolus. The MEP peak-to-peak amplitudes will be measured from left and right tibialis anterior and abductor hallucis muscles. Stimulation parameters will be varied in order to achieve the maximum amplitude values. Evoked potentials will be measured before and at 10 and 30 minutes after the start of the magnesium infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Crawford, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada